CLINICAL TRIAL: NCT07200063
Title: Comparative Assessment of Children's Acceptance and Compliance of Mouthwash Containing Silver Nanoparticles Compared to Chlorhexidine Mouthwash: A Randomized Clinical Trial.
Brief Title: Children Acceptance of AgNP Mouthwash Against Chlorhexidine Mouthwash
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahem Mohamed Ibrahem Arafat, Master's student (Dentist), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AgNP vs CHX Mouthwashes
Record Dates: First submitted 2025-09-09; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Teeth Staining; Numbness of the Tongue and Soft Tissue; Bitter Taste
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: randomized clinical trail on three groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- use AgNP mouthwash as experimental group (Experimental): nano cure mouthwash
  Interventions: Other: nano silver mouthwash
- use hexitol mouthwash (CHX) as experimental group (Experimental)
  Interventions: Other: Chlorhexidine mouthwash (0.12%)
- orovex mouthwash (CHX) as a comparator group (Active Comparator)
  Interventions: Other: Chlorhexidine mouthwash (0.2%)

INTERVENTIONS:
Other: nano silver mouthwash — nano silver mouthwash will reduce the side effect of chlorhexidine and increase acceptance of the mouthwash to patients
  Arms: use AgNP mouthwash as experimental group
Other: Chlorhexidine mouthwash (0.12%) — the concentration of chlorhexidine
  Arms: use hexitol mouthwash (CHX) as experimental group
Other: Chlorhexidine mouthwash (0.2%) — chlorhexidine mouthwash 0.2% (orovex )
  Other Names: orovex
  Arms: orovex mouthwash (CHX) as a comparator group

SUMMARY:
This study aims to evaluate and compare the children's acceptance of mouthwash containing silver nanoparticles versus Chlorhexidine.

DETAILED DESCRIPTION:
Effective management of dental plaque is crucial for preventing periodontal diseases, dental caries, and other oral health complications. Oral hygiene can be maintained through both chemical and mechanical methods. Chemical methods are particularly beneficial in situations where mechanical cleaning proves challenging. Mouthwashes represent a significant chemical strategy for controlling plaque. Among different types of mouthwashes, chlorhexidine is considered the gold standard due to its high efficacy against a broad spectrum of bacteria and its role in plaque management, which helps prevent periodontal diseases. However, it is important to note that chlorhexidine has several side effects, such as numbness, changes in taste perception, dental staining, and an unpleasant bitter taste.

In modern applications, nanotechnology is being utilized more frequently, especially with the integration of nanoparticle materials. Silver nanoparticles, in particular, are widely used in the medical field because of their remarkable antibacterial effects on oral biofilms associated with periodontal disease.

Therefore, this research aims to evaluate the children's acceptance of chlorhexidine mouthwash in children compared to a mouthwash containing silver nanoparticles, as well as to assess their respective impacts on gingivitis.

ELIGIBILITY:
Inclusion criteria

* Children aged from 6 to 12 in good general health and medically free
* Cooperative patient who will care about attending the follow-up visit
* Acceptance of the parents to sign the informed consent
* Composite restoration on anterior teeth Exclusion criteria
* Children who are unable to attend the follow-up visit
* Medically compromised patient
* Handi-capped patient
* Parents refuse to sign informed consent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
children acceptance and compliance | 15 days
  it will be measured by likert scale (1-5)
  1 (strongly disagree) 5 (strongly agree)

SECONDARY OUTCOMES:
Gingival health | 15 days
  * gingival inflammation measured by modified gingival index scoring criteria (0-4) 0 (Normal gingiva ) 4 (sever inflammation of gingiva)
plaque thickness at gingival margin | 15 days
  * measure plaque thickness at gingival margin by plaque index by loe and silness scoring criteria (0-3) 0 (no plaque) 3 (thick plaque)
color stability of composite restoration of anterior teeth | 15 days
  measure color stability of composite restoration of anterior teeth ΔE* = √((L₂ - L₁)² + (a₂ - a₁)² + (b₂ - b₁)²
  Where:
  L* = Lightness (0 = black, 100 = white)
  1. = Red-Green axis (positive = red, negative = green)
  2. = Yellow-Blue axis (positive = yellow, negative = blue
     * L1, a1, b1 = before exposure
     * L2, a2, b2 = after exposure A higher ∆E means more discoloration.

IPD SHARING:
Plan to Share IPD: No
cause it a private data and it's mentioned in the informed consent that the data of the participants will be private and not published